CLINICAL TRIAL: NCT03341468
Title: Use of a Urethral Catheter Immobilization Device to Reduce Pain and Discomfort Associated With Catheter Mobility in Post-Prostatectomy Patients
Brief Title: Urethral Catheter Immobilization Device to Reduce Catheter-Related Discomfort
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI confirmed no subjects consented and stated study not started due to insufficient staffing and once staff on board, the COVID-19 public health emergency occurred.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Shahin Tabatabaei, Assistant Professor of Urology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017P001343
Record Dates: First submitted 2017-10-16; First posted 2017-11-14 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Urinary Catheter-Related Discomfort
Keywords: Urethral catheter discomfort; Urethral catheter pain; Urethral catheter immobilization device; Prolonged urethral catheterization; Foley catheter; Urinary catheter; Indwelling urethral catheter support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Urethral catheter immobilization (Experimental): Subjects randomized to the intervention group will undergo radical prostatectomy with placement of the urethral catheter per the standard of care. The urethral catheter immobilization device will be applied in the operating room prior to the patient being transported to the recovery room. Subjects will be informed on safe use of the device and must demonstrate competency in removing and replacing the device prior to discharge. Subjects will also be given an elastic leg strap, which they may use concurrently with the device. Subjects will attend routine follow up appointments with their surgeon for removal of the urethral catheter and void trial per standard of care, at which the device will no longer be needed.
  Interventions: Device: Urethral catheter immobilization
- No urethral catheter immobilization (No Intervention): Subjects randomized to the control group will undergo radical prostatectomy with placement and securing of the urethral catheter per the standard of care. The catheter will be secured to the leg using cloth tape. Subjects will also be given an elastic leg strap that they may use following discharge, as is routine. Subjects will attend routine follow up appointments with their surgeon for removal of the urethral catheter and void trial per standard of care.

INTERVENTIONS:
Device: Urethral catheter immobilization — Subjects assigned to the control group will undergo radical prostatectomy with placement and securing of the urethral catheter per the standard of care. The catheter will be secured to the leg using cloth tape. Subjects will also be given an elastic leg strap that they may use following discharge, as is routine. Subjects will attend routine follow up appointments with their surgeon for removal of the urethral catheter and void trial.
  Subjects will be asked to fill out a symptom-based questionnaire prior to leaving the office. This will conclude their participation in the study.
  Other Names: Indwelling urethral catheter support
  Arms: Urethral catheter immobilization

SUMMARY:
This is a randomized controlled study to determine the efficacy and safety of a patented urethral catheter support device designed to reduce discomfort associated with urethral catheter mobility in males.

Movement of a catheter within the urethra is a source of discomfort for patients. The investigators hypothesize that this discomfort can be reduced by using an external device designed to securely fasten the catheter to the penis.

DETAILED DESCRIPTION:
Indwelling urethral catheters are a source of discomfort and pain in males, particularly when in place for extended periods of time. All patients require catheterization for a minimum of 10 days following radical prostatectomy. Currently, catheters are secured to the patient's leg using tape or an elastic leg strap. This point of securing, however, allows the tip of the penis and the urethral meatus to move in different vectors from the catheter. Data demonstrating urethral catheter hypermobility as an etiology of pain and discomfort have not been reported. However, clinical experience suggests that this type of catheter mobility is associated with significant discomfort.

It is predicted that the use of an external urethral catheter immobilization device (Patent: Simpson et al., US8500719, 2013) designed to secure/minimize catheter movement relative to the tip of the penis will greatly improve catheter associated pain and discomfort in men undergoing radical prostatectomy. The catheter immobilization device is an FDA-approved, 510(k) exempt, pliant tubular structure comprised of Suprazote Foam (Zotefoams) that surrounds the penile shaft. The foam support has a rigidity greater than that of the flaccid penis. It is bi- lobed (i.e., two identical halves) that hinge together to close around the tip of the penis with an aperture aligned with the urethra. The catheter extends through this opening and is secured to the device does not alter the urethral catheter in any fashion. The device limits catheter movement radial to the axis of the catheter. This, in turn, keeps the catheter in line with the urethra, reducing abrasion and traction to the meatus and urethra.

To test the hypothesis, a randomized-controlled trial will be performed in male patients who underwent radical prostatectomy. These men will be randomized to two arms: one arm will have the device fitted around their catheter after surgery is complete while the other will not have the device fitted. Outcome measures involving catheter-related pain and discomfort will then be assessed until the urethral catheter is removed per standard of care after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo radical prostatectomy at the Massachusetts General Hospital
* Anticipated intra-operative placement of an 18 or 20 French, latex or silicone urethral catheter at the conclusion of the operation (standard of care)
* At least 18 years of age

Exclusion Criteria:

* Inability to speak, read or understand English
* Apparent sore, rash, or infection on the penis
* Anatomic abnormalities that would prevent proper application and use of the device
* Patients with significant physical or mental disability that, in the opinion of the treating surgeon, might prevent safe placement or removal of the device, or completion of the symptom-based survey.
* Patients with fragile skin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Urethral catheter related pain/discomfort | At follow-up visit for foley removal (10 days after surgery)
  To be assessed via a proprietary questionnaire that is multiple choice and designed to determine the nature of catheter related pain/discomfort. Pain is to be measured on a scale of 1 to 10. Subsequent descriptions of the pain (location, aggravating factors, relieving factors, etc.) and impact are to be answered as multiple choice questions so as to structure the responses without limiting the response.

SECONDARY OUTCOMES:
Adverse events secondary to urethral immobilization | Through post-operative day # 1 and at follow-up visit for foley removal (10 days after surgery)
  Complications related to the urethral catheterization immobilization device will be assessed including pain/discomfort related to the device itself, urinary tract infection, skin rash, compromised skin integrity, skin infection, penile edema, restricted blood flow to penis, penile necrosis secondary to restricted blood flow, tightness or discomfort during erection, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Tabatabaei, MD, Principal Investigator — Massachusetts General Hospital, Department of Urology
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No